CLINICAL TRIAL: NCT06892873
Title: Clinical Evaluation and Comparison of Pain Acceptance of Different Types of Injection Systems in Palatal Anesthesia Applied to Children
Brief Title: Clinical Evaluation and Comparison of Pain Acceptance of Different Types of Injection Systems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Halenur Altan, Associate Professor, Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NecmettinEU04
Record Dates: First submitted 2024-11-29; First posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Dental Anesthesia
Keywords: Dental Anxiety; Jet Injection; Dental Injection; Pain Assessment; Palatal Infiltration Anesthesia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Application of Traditional Dental Injection Method (Active Comparator): Conventional dental injection was applied.
  Interventions: Other: Traditional dental injection
- Application of Comfort-in Jet Injection Method (Experimental): Comfort-in Jet injection was applied.
  Interventions: Device: Comfort-In

INTERVENTIONS:
Device: Comfort-In — Application of Comfort-in Jet Injection Method Comfort-in jet injection method was used for palatal anesthesia of the primary molars. The device was placed 5 mm below the palatal gingival margin, close to the free gingiva, and with a steep angle. 0.2 ml of anesthetic solution was administered by pressing the jet injection system button. 1 mL Articaine Hydrochloride (Ultracaine D-S forte, Hoechst, Canada) containing 1/100,000 epinephrine was used as a local anesthetic agent in the injections. 38 patients were included in this group and the procedure was performed. After waiting for 2 minutes, the anesthetized area was probed with the help of a probe (probing gingiva) to check whether the anesthesia had taken effect. Afterwards, buccal infiltration anesthesia was performed with the help of a traditional dental injector and tooth extraction was performed.
  Arms: Application of Comfort-in Jet Injection Method
Other: Traditional dental injection — Application of Traditional Dental Injection Method Palatal injection; It was applied 5-10 mm below the palatal gingival margin*, on the attached gum, and with a 45-degree needle angle. After needle entry, 0.2 mL of anesthetic solution was stored when bone contact was removed. 1 mL Articaine Hydrochloride (Ultracaine D-S forte, Hoechst, Canada) containing 1/100,000 epinephrine and a 27 G dental needle were used as local anesthetic agents for injections. 38 patients were included in this group and the procedure was performed. After waiting for 2 minutes, the anesthetized area was probed with the help of a probe (probing gingiva) to check whether the anesthesia had taken effect. Afterwards, buccal infiltration anesthesia was performed with the help of a traditional dental injector and tooth extraction was performed.
  Arms: Application of Traditional Dental Injection Method

SUMMARY:
The goal of this randomized clinical trial is to compare two different injection methods in children. The main question it aims to answer is:

Is the needle-free injection method more painless than the traditional dental method?

Two different methods will be used for children to perform anesthesia for extraction permanent molars.

DETAILED DESCRIPTION:
The reason for wanting to conduct this research is that palatal injection, which is routinely used in the extraction of primary molars, causes pain and fear due to the tight connection between the palatal mucosa and the bone, and causes difficulty in tolerating it by pediatric patients. The aim of our research is to evaluate whether Comfort-in™ Needle-Free Injection, which can be used during palatal injection, can reduce injection pain. The palate side of the upper primary molars that require extraction treatment will be anesthetized with two different anesthesia techniques. One of these techniques will be applied with a needle and the other without a needle. The technique will be decided by determining which technique will be applied first using a random computer program. A 'popcorn sound' may occur during needle-free anesthesia, the investigators wanted to inform participants in advance so that participants are not surprised. The investigators also want to apply a scale called IDAF-4C to participants in order to learn the level of participants' concerns and fears about dentistry. The investigators plan to ask participants about this scale when participants first come to the clinic. After anesthetizing participants' teeth, the investigators will ask participants to evaluate the severity of pain with the Wong-Baker Pain Rating Scale. During female anesthesia, body responses will be recorded via video and then evaluated with the FLACC scale.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 4-11 years
* Bilateral maxillary primary molars with an indication for extraction
* Not having taken any analgesics up to 12 hours before treatment
* Not having used antibiotics in the last month
* Teeth with at most 1/2 of the root physiologically resorbed
* Systemically healthy children
* Those who agreed to participate in the study
* Those who scored 1-2-3-4 according to the Frankl behavior scale
* Frankl 1: Patients who refuse treatment, cry, are extremely fearful or show signs of severe negative behavior
* Frankl 2: Patients who are noncompliant, unwilling to receive treatment, show signs of unclear negative behavior, are sullen but do not express anxiety
* Frankl 3: Patients who accept treatment, are compliant, shy, establish a relationship with the physician but approach it moderately
* Frankl 4: Patients who cooperate with the physician, are curious about the treatment, smile and are happy with the environment (Frankl 1962)

Exclusion Criteria:

* If the infection has not spread beyond 1/3 of the root or furcation area
* If the root formation of the permanent tooth below is not complete or 2/3 root formation is not formed
* In the presence of dentigerous or follicular cysts
* Teeth with excessive material loss
* Teeth without permanent tooth germ underneath
* Teeth with suspected malignancy
* Children who are not systemically healthy
* Patients with a previous history of allergy to local anesthetics
* If the teeth to be extracted will require surgical extraction during the procedure
* Acute infection status (clinically, the patient has any systemic findings such as mild or severe pain, swelling, trismus, fever, lymphadenopathy, weakness, headache or nausea)
* Those who do not accept to participate in the study

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 76 (Actual)
Dates: Start 2024-01-22 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-09-06 (Actual)

PRIMARY OUTCOMES:
Pain Perception of Wong-Baker Scale | 1 minute after anesthesia application, the patient is asked to score the pain they feel.
  The investigators expect the comfort-in jet injection method to produce a lower score on the Wong-Baker pain scale than the traditional anesthesia method.The Wong-Baker pain scale is scored between 0-10. 0 means the patient has no pain and 10 means they feel very severe pain.
Pain Perception of The Face, Legs, Activity, Cry, and Consolability (FLACC) scale | The video was taken to examine the patient's body reactions during application of the anesthesia method. The data were evaluated up to 2 day.
  The investigators expect the comfort-in jet injection method to produce a lower score on the FLACC scale applied to pain acceptance in pediatric patients compared to the traditional anesthesia method. The FLACC pain scale is scored between 0-10. 0 means that the patients pain acceptance is good and 10 means that the pain acceptance is low.
Evaluation of physiological parameters with Pulse Oximetry | Data were recorded during applying anesthesia. Data were evaluated for up to 2 days.
  A finger-type pulse oximeter was used to measure pulse and oxygen saturation values. Data were recorded before and after anesthesia.

CONTACTS AND LOCATIONS:
Overall Officials: Halenur Altan, Principal Investigator — halenuronat@gmail.com
Locations (1):
- Necmettin Erbakan University, Faculty of Dentistry, Konya, Meram, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Altan H, Belevcikli M, Cosgun A, Demir O. Comparative evaluation of pain perception with a new needle-free system and dental needle method in children: a randomized clinical trial. BMC Anesthesiol. 2021 Dec 1;21(1):301. doi: 10.1186/s12871-021-01524-1. PMID 34852779

DOCUMENTS (1):
  • Study Protocol (2023-12-08): https://cdn.clinicaltrials.gov/large-docs/73/NCT06892873/Prot_000.pdf